CLINICAL TRIAL: NCT01212146
Title: A Randomized Double-blind, Crossover Clinical Trial to Assess the Efficacy of Lactobacillus Paracasei Enriched Artichokes in the Treatment of Functional Constipation
Brief Title: Probiotic-enriched Artichoke in Functional Constipation
Acronym: PAFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Francesco Russo, MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0818G
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Functional Constipation
Keywords: Artichokes; Constipation; Functional Foods; Prebiotics; Probiotics
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic-enriched Artichokes (Experimental): Artichokes containing approximately 1.20 x 10^8 CFU of live probiotic cells of Lactobacillus paracasei IMPC 2.1 LMGP22043 per gramme
  Interventions: Dietary Supplement: Lactobacillus paracasei IMPC 2.1 LMGP22043
- Ordinary artichokes (Active Comparator): Ordinary artichokes (probiotic free) of identical shape, texture, and appearance of probiotic-enriched artichokes
  Interventions: Dietary Supplement: Ordinary artichokes

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei IMPC 2.1 LMGP22043 — participants will complement their usual lifestyles and dietary intakes with probiotic artichokes, enriched with the probiotic strain Lactobacillus paracasei IMPC2.1 (LMGP22043). The product contains approximately 1.20 x 10^8 CFU of live probiotic cells of Lactobacillus paracasei IMPC 2.1 LMGP22043 per gramme, which resulted in a daily dose of about 2 x 10^10 CFU.
  Arms: Probiotic-enriched Artichokes
Dietary Supplement: Ordinary artichokes — Probiotic artichokes will be tested against ordinary artichokes (probiotic free) of identical shape, texture, and appearance produced by the same manufacturer. Artichokes will be put in similar packages and there will be no way to distinguish between the two products.
  Arms: Ordinary artichokes

SUMMARY:
The aim of the present randomized double-blind controlled crossover study is to compare the effects of the 15-day consumption of artichokes enriched with the probiotic Lactobacillus paracasei LMGP22043 with those of ordinary artichokes on treatment preference, satisfactory relief of symptoms, bowel habit and the modulation of SCFA production in a group of patients suffering from functional constipation.

DETAILED DESCRIPTION:
Functional constipation is a common problem in westernized societies and is characterized by different gastrointestinal symptoms.Different therapeutic strategies have been proposed, but a new therapeutic approach for constipation could be based on the modulation of intestinal microflora by administering prebiotics and/or probiotics. Currently, probiotic products are mainly incorporated in fermented milk-based products or concentrated probiotic preparations. To enlarge the range of choice and to exploit the nutritional qualities of plant matrices, an innovative line of probiotic vegetable products such as artichokes has been developed. The use of these vegetables containing live probiotic strains can take advantage of some their peculiar features for growth and improved bacterial survival. Artichokes can, therefore, work as valid "active" vehicles for the transport and release of adequate amounts of bacterial populations.

ELIGIBILITY:
Inclusion Criteria:

* fulfilment of the Rome Criteria III for constipation
* availability of at least one GI imaging study during the last five years(colonoscopy, sigmoidoscopy, abdominal ultrasound, barium enema)
* commitment to availability for the whole study period

Exclusion Criteria:

* major abdominal surgery
* the presence of any concomitant diseases such as organic GI diseases including lactose and gluten intolerance; medical or psychiatric illness
* alarming symptoms (rectal bleeding, weight loss, etc)
* family history of peptic ulcer, colorectal cancer, or IBD;
* abnormal laboratory data or thyroid function.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Treatment preference | After treatment with artichokes enriched with probiotics (period 1: 15 days) and at the end of treatment with ordinary artichokes (period 2: 15 days)
  The participants will be asked about treatment preference (the period with least symptoms) at the last visit.

SECONDARY OUTCOMES:
Visual analogue score (VAS) of satisfactory relief of symptoms | At the end of the run-in period (7 days), after treatment with artichokes enriched with probiotics (period 1: 15 days) and at the end of treatment with ordinary artichokes (period 2: 15 days)
  The participants will be asked about satisfactory relief of symptoms by using a visual analogue scale (VAS) with grades from 0 (no relief) to 100 (best imaginable relief of symptoms). VAS values will be categorized in 4 classes: 0-25: no or poor relief of symptoms, 26-50: moderate relief of symptoms; 51-75: good relief of symptoms; 76-100: very good relief of symptoms.
GSRS sum score | At the end of the run-in period (7 days), after treatment with artichokes enriched with probiotics (period 1: 15 days) and at the end of treatment with ordinary artichokes (period 2: 15 days)
  The GSRS (Gastrointestinal Symptom Scoring Rate) is a validated questionnaire for GI symptoms. GSRS utilizes a seven-level Likert scale (1 to 7), depending on intensity and frequency of GI symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Riezzo, MD, Study Director — National Institute of Digestive Diseases IRCCS "S. de Bellis"
Locations (1):
- National Institute for Digestive Diseases IRCCS "S. de Bellis", Castellana Grotte, Bari, Italy

REFERENCES:
- [Background] Higgins PD, Johanson JF. Epidemiology of constipation in North America: a systematic review. Am J Gastroenterol. 2004 Apr;99(4):750-9. doi: 10.1111/j.1572-0241.2004.04114.x. PMID 15089911
- [Background] Kleessen B, Schwarz S, Boehm A, Fuhrmann H, Richter A, Henle T, Krueger M. Jerusalem artichoke and chicory inulin in bakery products affect faecal microbiota of healthy volunteers. Br J Nutr. 2007 Sep;98(3):540-9. doi: 10.1017/S0007114507730751. Epub 2007 Apr 20. PMID 17445348
- [Background] Valerio F, De Bellis P, Lonigro SL, Morelli L, Visconti A, Lavermicocca P. In vitro and in vivo survival and transit tolerance of potentially probiotic strains carried by artichokes in the gastrointestinal tract. Appl Environ Microbiol. 2006 Apr;72(4):3042-5. doi: 10.1128/AEM.72.4.3042-3045.2006. PMID 16598015
- [Derived] Riezzo G, Orlando A, D'Attoma B, Guerra V, Valerio F, Lavermicocca P, De Candia S, Russo F. Randomised clinical trial: efficacy of Lactobacillus paracasei-enriched artichokes in the treatment of patients with functional constipation--a double-blind, controlled, crossover study. Aliment Pharmacol Ther. 2012 Feb;35(4):441-50. doi: 10.1111/j.1365-2036.2011.04970.x. Epub 2012 Jan 8. PMID 22225544